CLINICAL TRIAL: NCT06460402
Title: Comparing Ice Therapy and Warm Baths for Hemorrhoidectomy Wound Care
Brief Title: Ice Therapy and Warm Baths for Hemorrhoidectomy Wound Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMRP23113N
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Post Hemorrhoidectomy Pain; Post Operative Pain; Wound Heal
Keywords: pain; hemorrhoids
MeSH Terms: conditions — Pain, Postoperative; Pain; Hemorrhoids

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-group controlled trial comparing the effects of cryotherapy versus warm water sitz baths on post-hemorrhoidectomy wound care. Eligible participants (N=128) will be 1:1 randomized to receive either ice pack applications (cryotherapy group) or warm water sitz baths (control group) after undergoing surgical hemorrhoid excision. The primary outcomes of postoperative pain levels and analgesic consumption, as well as secondary outcomes of wound separation incidence and swelling, will be assessed at various time points. This parallel-group design allows direct comparison of the two interventions to determine if cryotherapy is superior to the current standard of care (sitz baths) in promoting recovery after hemorrhoidectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice packing (Experimental): Participants in this arm will receive cryotherapy in the form of ice pack applications to the perianal area for 20 minutes every 2 hours during the first 48 hours after hemorrhoidectomy. The ice packs will be applied externally to the surgical site to reduce pain, swelling, and inflammation. Participants will be instructed on proper ice pack application techniques and will be provided with the necessary supplies. Postoperative pain levels, analgesic consumption, wound healing, and other outcomes will be assessed at various time points.
  Interventions: Other: Ice packing
- Warm sitz bath (Active Comparator): Participants in this arm will receive warm water sitz baths as the standard postoperative care after hemorrhoidectomy. They will be instructed to sit in a bathtub or a special sitz bath basin filled with warm water for 15-20 minutes, 2-3 times daily, starting from the first postoperative day. The warm water is believed to promote blood flow, relax the anal sphincter, and soothe the perianal area, potentially aiding in pain relief and wound healing. Participants will be provided with instructions on proper sitz bath techniques and will be assessed for postoperative pain, analgesic consumption, wound healing, and other outcomes at various time points, similar to the cryotherapy arm.
  Interventions: Other: Warm sitz bath

INTERVENTIONS:
Other: Ice packing — For both arms, participants will self-administer interventions at home per instructions: ice packs every 2 hours for 48 hours (ice pack arm) or sitz baths 2-3 times daily for 7 days (warm water arm). Standardized supplies and daily logs will be provided. All participants receive standard postop care with analgesics and wound care. Adverse events will be monitored closely. Intervention duration: 48 hours (ice), 7 days (sitz bath). Assessments: baseline, 24/48/72 hours (pain, swelling), 1 week (wound separation). Total study duration per participant: ~1 week from surgery.
  Arms: Ice packing
Other: Warm sitz bath — Participants in this arm will receive standard instructions to perform warm water sitz baths at home, starting from the day of surgery and continuing for 7 days postoperatively. They will be advised to take 2-3 sitz baths per day, with each bath lasting for 15-20 minutes. A standard plastic sitz bath basin will be provided to the participants, along with a thermometer to monitor the water temperature. The recommended water temperature range for the sitz baths is 37-40°C (98.6-104°F). Participants will be instructed to keep a daily log recording the number of sitz baths taken, the duration of each bath, and the water temperature. Proper hygiene and wound care instructions will also be provided to prevent infection.
  Arms: Warm sitz bath

SUMMARY:
This study aims to compare the effectiveness of cryotherapy and warm water sitz bath in post-hemorrhoidectomy wound care. It is a prospective, randomized controlled trial that will assess the impact of these two methods on postoperative pain, analgesic use, wound separation, and swelling.

DETAILED DESCRIPTION:
Background: Hemorrhoids are a common anorectal condition. For patients with severe or intolerable symptoms, surgical excision (hemorrhoidectomy) is an effective treatment. However, postoperative pain, swelling, and wound complications are common issues that may delay recovery. Currently, warm water sitz baths are recommended for pain relief and healing, but some studies suggest cryotherapy may be an effective alternative by reducing inflammation and swelling. This trial aims to systematically compare the effects of these two therapies.

Objectives:

Primary: Assess and compare pain levels (VAS) and total analgesic consumption between the two groups at different postoperative time points.

Secondary: Evaluate and compare wound separation incidence at 1-week follow-up and wound swelling at different time points.

Methods:

Design: Prospective, randomized, parallel-controlled trial with 1:1 allocation. Subjects: 128 symptomatic hemorrhoid patients (18-75 years old) undergoing hemorrhoidectomy, randomized into cryotherapy or sitz bath group.

Intervention: Cryotherapy group - ice packs for 20 min every 2h within 48h post-op. Sitz bath group - warm water baths 2-3 times daily for 15-20 min.

Outcome measures: Pain VAS scores, analgesic consumption, wound separation rate, swelling assessment at different time points.

Expected results and benefits: Cryotherapy is hypothesized to result in lower pain scores, reduced analgesic use, lower wound separation incidence and milder swelling compared to sitz baths. This may lead to improved postoperative recovery and quality of life for patients.

Risks and management: Potential mild adverse reactions like skin irritation, temporary nerve stimulation will be closely monitored and appropriately managed. The study will be terminated for any severe adverse events.

Statistical analysis: Repeated measures ANOVA for VAS scores and analgesic use. Chi-square or Fisher's exact test for wound separation rates. Descriptive statistics for baseline characteristics.

In summary, this well-designed randomized control trial aims to provide high-quality evidence comparing cryotherapy and sitz baths in post-hemorrhoidectomy care, potentially identifying a superior treatment option to improve patient outcomes and experiences.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years Diagnosed with symptomatic hemorrhoids requiring surgical removal Able to understand and comply with the trial procedures

Exclusion Criteria:

Pregnant or lactating women Known allergy to cold or warm therapy Coagulation disorders or receiving anticoagulant therapy Severe organ dysfunction (cardiac, pulmonary, hepatic, renal, etc.) Immunocompromised or receiving immunosuppressive therapy Other anorectal surgery within the past 1 month Concomitant anorectal diseases (e.g., anal fistula, anal fissure) requiring additional surgical treatment Cognitive impairment, psychiatric illness, or language barrier preventing compliance Currently participating in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores | at 24, 48, and 72 hours post-surgery for pain.
  Pain scores assessed using the Visual Analog Scale (VAS) at 24, 48, and 72 hours after hemorrhoidectomy surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- E-Da hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data from this clinical trial with other researchers. All participant data will remain confidential and will only be used for the purposes of this specific study by the research team at E-DA hospital

REFERENCES:
- [Derived] Chen PC, Kao YK, Yang PW, Chen CH, Chen CI. Ice Packing Versus Warm Sitz Baths for Post-hemorrhoidectomy Pain Management: A Randomized Controlled Trial. Dis Colon Rectum. 2025 Jul 1;68(7):865-874. doi: 10.1097/DCR.0000000000003707. Epub 2025 Mar 27. PMID 40145987